CLINICAL TRIAL: NCT02680158
Title: A Randomized, Controlled, Double-Masked, Multicenter Trial Designed to Evaluate Acute Tear Production With the Oculeve Intranasal Lacrimal Stimulator Compared to Two Control Applications in Patients With Aqueous Deficient Dry Eye
Brief Title: A Study to Evaluate the Safety and Effectiveness of Oculeve Intranasal Lacrimal Neurostimulator in Participants With Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: OCUN-009
Record Dates: First submitted 2016-01-21; First posted 2016-02-11 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndrome; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Three way cross-over study with 6 sequences.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Sequence 1-Intranasal: Extranasal: Sham (Experimental): Oculeve device, intranasal (test) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by sham device, intranasal (control) application, for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal
- Sequence 2-Intranasal: Sham: Extranasal (Experimental): Oculeve device, intranasal (test) application for approximately 3 minutes followed by sham device, intranasal (control) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal
- Sequence 3-Extranasal: Intranasal: Sham (Experimental): Oculeve device, extranasal (control) application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes, followed by sham device (control), intranasal application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal
- Sequence 4-Extranasal: Sham: Intranasal (Experimental): Oculeve device, extranasal (control) application for approximately 3 minutes followed by sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal
- Sequence 5-Sham: Intranasal: Extranasal (Experimental): Sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal
- Sequence 6-Sham: Extranasal: Intranasal (Experimental): Sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes followed by on Day 0. There was rest period of 60 minutes before proceeding to the next application.
  Interventions: Device: Oculeve Intranasal; Device: Sham; Device: Oculeve Extranasal

INTERVENTIONS:
Device: Oculeve Intranasal — Oculeve device, intranasal (test) application for approximately 3 minutes.
Device: Sham — Sham device (control), intranasal application for approximately 3 minutes.
Device: Oculeve Extranasal — Oculeve device, extranasal (control) application for approximately 3 minutes.

SUMMARY:
The purpose of this study is to compare acute tear production produced by the Oculeve Intranasal Lacrimal Neurostimulator with two control devices in participants with aqueous tear deficiency.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, double-masked, multicenter clinical trial in which participants with aqueous tear deficiency will receive three different device applications in a randomized sequence.

ELIGIBILITY:
Inclusion Criteria:

* Participants with aqueous tear deficiency
* Literate, able to speak English or Spanish, and able to complete questionnaires independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol

Exclusion Criteria:

* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to clinically significant increased bleeding
* Nasal or sinus surgery including nasal cautery or significant trauma
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Diagnosis of epilepsy
* Corneal transplant in either or both eyes
* Participation in any clinical trial with a new active substance or a new device within 30 days of the Screening Visit
* A woman who is pregnant, planning a pregnancy, or nursing at the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Study Director — Allergan
Locations (2):
- United States (2):
  - The Eye Care Group, Waterbury, Connecticut
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sheppard JD, Torkildsen GL, Geffin JA, Dao J, Evans DG, Ousler GW, Wilson J, Baba SN, Senchyna M, Holland EJ. Characterization of tear production in subjects with dry eye disease during intranasal tear neurostimulation: Results from two pivotal clinical trials. Ocul Surf. 2019 Jan;17(1):142-150. doi: 10.1016/j.jtos.2018.11.009. Epub 2018 Nov 22. PMID 30472141

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Sequence 1 - Intranasal : Extranasal : Sham: Oculeve device, intranasal (test) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by sham device, intranasal (control) application, for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
- Sequence 2 - Intranasal : Sham : Extranasal: Oculeve device, intranasal (test) application for approximately 3 minutes followed by sham device, intranasal (control) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
- Sequence 3 - Extranasal: Intranasal: Sham: Oculeve device, extranasal (control) application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes, followed by sham device (control), intranasal application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
- Sequence 4 - Extranasal : Sham : Intranasal: Oculeve device, extranasal (control) application for approximately 3 minutes followed by sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes on Day 0. There was rest period of 60 minutes before proceeding to the next application.
- Sequence 5 - Sham : Intranasal : Extranasal: Sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by on Day 0. There was rest period of 60 minutes before proceeding to the next application.
- Sequence 6 - Sham : Extranasal : Intranasal: Sham device (control), intranasal application for approximately 3 minutes followed by oculeve device, extranasal (control) application for approximately 3 minutes followed by oculeve device, intranasal (test) application for approximately 3 minutes followed by on Day 0. There was rest period of 60 minutes before proceeding to the next application.
Period: Overall Study
Arm/Group | Sequence 1 - Intranasal : Extranasal : Sham | Sequence 2 - Intranasal : Sham : Extranasal | Sequence 3 - Extranasal: Intranasal: Sham | Sequence 4 - Extranasal : Sham : Intranasal | Sequence 5 - Sham : Intranasal : Extranasal | Sequence 6 - Sham : Extranasal : Intranasal
Started | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes
Completed | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes | 8; 8 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: All randomized participants who were exposed to study application.
Units Other Than Participants: eyes
Groups:
- All Study Participants: All participants who received oculeve device, intranasal (test) application, extranasal (control) and sham device, intranasal (control) application, for approximately 3 minutes on Day 0.
Arm/Group | All Study Participants
Number analyzed (Participants) | 48
Number analyzed (eyes) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Acute Stimulated Tear Production
Description: Stimulated acute tear production in the study eye at Day 0 as measured by the difference between the Schirmer test score during stimulation and the test score before stimulation (basal). The Schirmer strip is placed just under the eyelid and wicks up the tears. It measures tear production on a linear scale of 0-35 mm. The study eye was defined as the eye with the greatest increase in tear production with stimulation by the cotton swab at Visit 1/Screening or, if there was no difference in stimulated tear production, the eye with the lower basal Schirmer score at Visit 2/Day 0 was selected. If there was no difference for either measure, the right eye was used as the study eye.
Time Frame: Day 0 post-application
Population: The FAS population included all randomized participants who were exposed to study application.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Groups:
- Oculeve Intranasal: Oculeve device, intranasal (test) application for approximately 3 minutes on Day 0
- Sham: Sham device (control), intranasal application for approximately 3 minutes on Day 0
- Oculeve Extranasal: Oculeve device, extranasal (control) application for approximately 3 minutes on Day 0
Arm/Group | Oculeve Intranasal | Sham | Oculeve Extranasal
Number analyzed (Participants) | 48 | 48 | 48
Number analyzed (eyes) | 48 | 48 | 48
mm | 25.3 (10.70) | 9.2 (7.34) | 9.5 (8.15)

2. Primary Outcome: Percentage of Participants Who Experienced One or More Device-related Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs in participants, users or other persons it does not necessarily have to have a causal relationship with the investigational medical device. Device-related AEs were presented as ocular and non-ocular.
Time Frame: Day 0
Population: Safety population included all randomized participants who were exposed to study application.
Measure: Number; unit: percentage of participants
Units Other Than Participants: eyes
Arm/Group | Oculeve Intranasal | Sham | Oculeve Extranasal
Number analyzed (Participants) | 48 | 48 | 48
Number analyzed (eyes) | 48 | 48 | 48
percentage of participants
  Device-related AEs (Ocular) | 0 | 0 | 0
  Device-related AEs (Non-ocular) | 4.2 | 0 | 0

3. Other Pre Specified Outcome: Corrected Distance Visual Acuity
Time Frame: 1-Day
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Slit Lamp Biomicroscopy
Time Frame: 1-Day
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Pulse Rate
Time Frame: 1-Day
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Oxygen Saturation
Time Frame: 1-Day
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Blood Pressure
Time Frame: 1-Day
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0
Description: Safety population included all randomized participants who were exposed to study applications.
Arm/Group | Oculeve Intranasal | Sham | Oculeve Extranasal
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 4/48 | 0/48 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oculeve Intranasal (N=48) | Sham (N=48) | Oculeve Extranasal (N=48)
Slight transient lightheadedness (General disorders) | 1 | 0 | 0
Intermittent nose itching (General disorders) | 1 | 0 | 0
Exacerbation of hypertension (General disorders) | 1 | 0 | 0
Corneal abrasion (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.